CLINICAL TRIAL: NCT02344628
Title: Randomized Controlled Trial Comparing Efficacy of Single Dose Treatment of Yaws With 20mg/kg Versus 30mg/kg of Azithromycin
Brief Title: Comparison of Two Different Doses of Azithromycin for Treatment of Yaws
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: World Health Organization (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Kwame Nkrumah University of Science and Technology (Other); Barcelona Institute for Global Health (Other); Papua New Guinea Institute of Medical Research (Other Government); Ghana Health Services (Other Government); Noguchi Memorial Institute for Medical Research (Other); Papua New Guinea National Department of Health (Unknown); University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSHTM-8832
Record Dates: First submitted 2015-01-17; First posted 2015-01-26 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2016-10

CONDITIONS: Yaws
MeSH Terms: conditions — Yaws | interventions — Azithromycin

ARMS (2):
- AZT30 (Active Comparator): Single dose of azithromycin at a dose of 30mg/kg - max 2 Grams
  Interventions: Drug: Azithromycin
- AZT20 (Experimental): Single dose of azithromycin at a dose of 20mg/kg - max 1 Grams
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Comparison of two different dosing strategies for the treatment of yaws

SUMMARY:
The study will be a single blinded, randomized, controlled open label non-inferiority phase III, trial with two parallel groups, conducted in Ghana and Papua New Guinea (PNG). The ultimate goal is to establish if a 20mg/kg dose of azithromycin is as effective as a 30mg/kg dose in the treatment of yaws. Approximately 600 clinically and serologically diagnosed yaws patients will be included in the study. Patients will be randomized to receive treatment with the two antibiotic regimens as follow: (i) Regimen I (AZT20): Single oral dose of 20 mg/kg azithromycin (ii) Regimen II (AZT30): Single oral dose of 30 mg/kg azithromycin. The follow-up period of patients will be 6 months. Assessments before, during and after the antibiotic treatment will include full medical history, clinical assessment of the lesion and, laboratory investigations. The primary efficacy parameters are healing of the lesion at 4 weeks and a four-fold decline in RPR titre at 6 months after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 to 16 years
* Clinical lesion consistent with primary or secondary yaws -Primary ulcer or papilloma
* Dually-Positive Chembio DPP Syphilis Screen & Confirm
* Informed Consent and Assent (for children 12-16 years)

Exclusion Criteria:

1. Known allergy to azithromycin or macrolides.
2. Treatment with long-acting penicillin or alternative antibiotic with activity against T. pallidum within the last 3 months (ceftriaxone, azithromycin or doxycycline, amoxicillin).
3. Patients with current treatment with any drugs likely to interact with the study medication.
4. Patients who are unable to take oral medication or having gastrointestinal disease likely to interfere with drug absorption.
5. Patients who may not be able to comply with the requirements of the study protocol including follow up visits.
6. Patients who are not willing to give informed consent (patient and/or parent/legal representative), or who withdraw consent.

Ages: 6 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 583 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Mabey, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (7):
- Ghana (4):
  - School Based Recruitment, Ayensuanor District, Eastern Region
  - School Based Recruitment, Upper West Akyem, Eastern Region
  - School Based Recruitment, West Akyem District, Eastern Region
  - School Based Recruitment, Nkwanta North District, Volta Region
- Papua New Guinea (2):
  - Community Based Recruitment, Karkar District, Madang Province
  - Community Based Recruitment, Kavieng Subdistrict, New Ireland Province
- London School of Hygiene and Tropical Medicine, London, United Kingdom

REFERENCES:
- [Derived] Marks M, Mitja O, Bottomley C, Kwakye C, Houinei W, Bauri M, Adwere P, Abdulai AA, Dua F, Boateng L, Wangi J, Ohene SA, Wangnapi R, Simpson SV, Miag H, Addo KK, Basing LA, Danavall D, Chi KH, Pillay A, Ballard R, Solomon AW, Chen CY, Bieb SV, Adu-Sarkodie Y, Mabey DCW, Asiedu K; study team. Comparative efficacy of low-dose versus standard-dose azithromycin for patients with yaws: a randomised non-inferiority trial in Ghana and Papua New Guinea. Lancet Glob Health. 2018 Apr;6(4):e401-e410. doi: 10.1016/S2214-109X(18)30023-8. Epub 2018 Feb 16. PMID 29456191

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZT30 | AZT20
Started | 291 | 292
Completed | 200 (4/52 clinical data was available for 283. Serological data 6/12 for 212. Both were available for 200) | 206 (4/52 clinical data was available for 286. Serological data 6/12 for 218. Both were available for 206)
Not Completed | 91 | 86

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZT30 | AZT20 | Total
Number analyzed (Participants) | 291 | 292 | 583
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 10 [8 to 12] | 10 [8 to 12] | 10 [8 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 88 | 171
  Male | 208 | 204 | 412
Region of Enrollment [Number; unit: participants]
  Papua New Guinea | 92 | 91 | 183
  Ghana | 199 | 201 | 400

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical and Serological Cure
Description: Clinical resolution of skin lesion at 4 weeks and at least four-fold decline in Rapid Plasma Reagin titre or seroreversion at 6-month (compared to baseline) in T.pallidum subsp. pertenue Polymerase Chain Reaction-confirmed subjects with yaws.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AZT30 | AZT20
Number analyzed (Participants) | 81 | 76
Participants | 68 | 61

2. Secondary Outcome: Number of Participants With Clinical and Serological Cure in Latent Yaws
Description: Clinical resolution of skin lesion at 4 weeks and at least four-fold decline in Rapid Plasma Reagin titre or seroreversion at 6-month (compared to baseline) in T.pallidum subsp. pertenue Polymerase Chain Reaction-negative.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | AZT30 | AZT20
Number analyzed (Participants) | 125 | 124
Participants | 65 | 73

3. Secondary Outcome: Number of Participants With Adverse Events
Description: To compare the incidences and relative risk of all Adverse Events (AEs), including treatment-related AEs, Serious Adverse Events (SAEs) and grade 3-4 toxicity in patients treated with AZT20 and AZT30 regimens
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | AZT30 | AZT20
Number analyzed (Participants) | 291 | 292
Participants | 12 | 14

ADVERSE EVENTS:
Arm/Group | AZT30 | AZT20
Serious Adverse Events (participants affected / at risk) | 0/291 | 0/292
Other Adverse Events (participants affected / at risk) | 12/291 | 15/292
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZT30 (N=291) | AZT20 (N=292)
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 2 | 0
Itching (Skin and subcutaneous tissue disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No